CLINICAL TRIAL: NCT05364541
Title: MyoVista wavECG Clinical Evaluation: >=60 y/o Enrichment Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heart Test Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HS-CLINVAL-002
Record Dates: First submitted 2022-04-28; First posted 2022-05-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-02

CONDITIONS: Health Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- MyoVista wavECG (Other): Single arm - subjects meeting the inclusion, exclusion and screening criteria will receive a MyoVista wavECG and a trans-thoracic echocardiogram.
  Interventions: Device: MyoVista wavECG

INTERVENTIONS:
Device: MyoVista wavECG — A standard 12-Lead, multi-channel resting interpretive trans-thoracic electrocardiograph providing both a Glasgow Interpretive Analysis and unique MyoVista wavECG Information for the detection of Left Ventricular Diastolic Dysfunction.

SUMMARY:
This is a single-center, interventional, single arm clinical study of the MyoVista wavECG for the detection of LV relaxation abnormalities. The study will be conducted at a single investigational site within the United States. Study subjects will predominately be screened from among those who have been enrolled in prior registry studies by the institution.

DETAILED DESCRIPTION:
The study has a planned enrollment of at least 50 subjects to obtain approximately 40 subjects with a "normal" septal and lateral e' value on echocardiogram. The criteria defined as septal e'< 7 cm/s or lateral e'< 10 cm/s for relaxation abnormality based on ASE/AECVI guidelines will be used for the evaluation of LV diastolic function which is associated with abnormal relaxation in echocardiography. An independent Core Lab will verify all septal and lateral e' values on the site-acquired echocardiograms and these Core Lab measurements will serve as the ground truth standard with regard to the presence of LV relaxation abnormalities.

Analysis of data from a prior multi-center study has revealed good correlation between the MyoVista wavECG results and echocardiography for the presence of LV relaxation abnormalities. This current study (HS-CLINVAL-002) is intended to supplement data collected in prior and ongoing studies, namely HS-CLINVAL-001, by recruiting individuals who are >60 years old and who are anticipated to have normal echocardiogram results based on a screening of selected clinical characteristics. Subjects in this study will be invited to participate and receive non-standard-of-care echocardiograms and a study driven MyoVista test.

The study will continue to focus on LV relaxation abnormalities by gathering additional device validation data for the purposes of regulatory approval peer-reviewed publications. Echocardiograms of study subjects will be used to compare/validate the study findings.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >=60 years of age
* Subjects will predominately be recruited among those who are already enrolled in existing registry studies within the institution.
* The subject provides written informed consent using an Informed Consent Form that is reviewed and approved by the site's Institutional Review Board (IRB).
* Conventional ECG results show a sinus rhythm and no other contraindicated rhythm abnormalities (see exclusions below).

Exclusion Criteria:

* The subject has current acute coronary syndrome, decompensated heart failure or stroke
* The subject has received any prior cardiac interventions or surgical therapeutic procedures relating to cardiac abnormalities: valve replacement, pacemaker implantation, coronary artery bypass grafting (CABG), heart transplant, ablation, coronary stent placement, etc.
* Conventional ECG results indicating a lack of sinus rhythm and/or any other contraindicated rhythm abnormalities, including: active atrial fibrillation or atrial flutter, left anterior fascicular block, left and/or right bundle branch block
* The subject is pregnant at the time of the study testing
* The subject has chest deformities that interfere with accurate measurement of ECG (either conventional or wavECG)
* Subjects with central nervous system or musculoskeletal abnormalities that may interfere with accurate acquisition of ECG and/or echocardiogram measurements.
* The subject is enrolled in another clinical study that may interfere with MyoVista or echocardiogram measurements. Exceptions to this may be approved by HeartSciences.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | Baseline
  Sensitivity and specificity of the MyoVista for the classification of Low e' where a "positive" includes a MyoVista wavECG result of Positive and Highly Positive. The study result will be considered to have achieved the pre-specified performance criteria for success if the sensitivity is demonstrated to exceed 70% and the specificity is demonstrated to exceed 70%.

CONTACTS AND LOCATIONS:
Overall Officials: Partho Sengupta, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- University of Texas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No